CLINICAL TRIAL: NCT05787132
Title: Comparison of the Balance Board and Perceptual Motor Therapy in Children With Cerebral Palsy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/ 01347 Bakhtawar Samejo
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; GMFC IV; GMFC V; Balance board; Perceptual motor therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Masking Description: This will be single blinded study. The data will be coded and the analyst will also be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Balance Board Therapy) (Experimental): 30 minutes of Balance board therapy along with conventional physical therapy
  Interventions: Other: Balance Board therapy
- Group B (Perceptual Motor Therapy) (Experimental): 30 minutes of Perceptual Motor therapy along with conventional physical therapy
  Interventions: Other: Perceptual Motor therapy

INTERVENTIONS:
Other: Balance Board therapy — Balance board therapy will be performed. balance board therapy has been shown to improve the sitting balance in children with cerebral palsy
  Arms: Group A (Balance Board Therapy)
Other: Perceptual Motor therapy — Perceptual motor therapy will be performed, it has been shown to improve dynamic sitting in children with cerebral palsy.
  Arms: Group B (Perceptual Motor Therapy)

SUMMARY:
Various studies have worked on the sitting balance of cerebral palsy (CP) with Gross Motor Function Classification System (GMFCS) level I-III with a sample greater than 30, there is no data available to compare the effect of a balance board and perceptual motor therapy to improve sitting in GMFCS level IV and V with a sample greater than 30. This study will add the authenticity to literature with a large sample size and affect the severity of the condition.

DETAILED DESCRIPTION:
This study will compare the effect of balance board therapy and Perceptual motor therapy to improve sitting in children with Cerebral palsy. Previous studies have worked on the sitting balance of cerebral palsy (CP) with Gross Motor Function Classification System (GMFCS) level I-III with a sample greater than 30, there is no data available to compare the effect of a balance board and perceptual motor therapy to improve sitting in GMFC level IV and V with a sample greater than 30. This study will add the authenticity to literature with large sample size and affect the severity of the condition. In addition, the patients with diagnosed Cerebral Palsy with GMFCS levels IV and V will be benefited from this study; an exercise program will help them to improve their sitting ability. A total of 88 Cerebral palsy patients will be included by dividing them into two groups (A, B). 1 hour of exercise session will be performed three times per week for 12 weeks with a total of 36 sessions. Both groups will receive 30 minutes of conventional physical therapy. In addition, group A will receive balance board therapy in the remaining 30 minutes while Group B will receive Perceptual motor therapy in the remaining 30 minutes. Data will be collected at baseline, at 4 weeks, at 8 weeks and at 12 weeks after intervention from both groups. The sitting balance will be measured by using Gross Motor Function Measure Scale (GMFM 88) and Trunk Control Motor Scale (TCMS).

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with CP GMFC level IV and V
* Both Male/Female
* Participants with the age ranges from 1.5 years to 5 years

Exclusion Criteria:

* Patients diagnosed with GMFC level I, II and III
* Participants taking botulinum toxin
* Participants diagnosed with auditory and visual impairments
* Participants diagnosed with mental impairments/ unable to understand the commands
* Participants diagnosed with any other comorbid conditions like (obesity, cardiovascular impairments)
* Participants who are not willing to participate

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 88 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function Measure Scale (GMFM 88) | Baseline
  The GMFM is standardized tool for measuring the change in gross motor function in children with cerebral palsy. GMFM-88 is four-point ordinal scale (0-3) with 88 items categorized in to 5 dimensions such as: lying and rolling (17 items), sitting (20 items), crawling and kneeling (14 items), standing (13 items), and walking, running and jumping (24 items). the average score ranges from 0-100. Higher scores indicate better capacity. The GMFM-88 reliability values range from 0.87 to 0.99
Gross Motor Function Measure Scale (GMFM 88) | 4th week
  The GMFM is standardized tool for measuring the change in gross motor function in children with cerebral palsy. GMFM-88 is four-point ordinal scale (0-3) with 88 items categorized in to 5 dimensions such as: lying and rolling (17 items), sitting (20 items), crawling and kneeling (14 items), standing (13 items), and walking, running and jumping (24 items). the average score ranges from 0-100. Higher scores indicate better capacity. The GMFM-88 reliability values range from 0.87 to 0.99
Gross Motor Function Measure Scale (GMFM 88) | 8th week
  The GMFM is standardized tool for measuring the change in gross motor function in children with cerebral palsy. GMFM-88 is four-point ordinal scale (0-3) with 88 items categorized in to 5 dimensions such as: lying and rolling (17 items), sitting (20 items), crawling and kneeling (14 items), standing (13 items), and walking, running and jumping (24 items). the average score ranges from 0-100. Higher scores indicate better capacity. The GMFM-88 reliability values range from 0.87 to 0.99
Gross Motor Function Measure Scale (GMFM 88) | 12th week
  The GMFM is standardized tool for measuring the change in gross motor function in children with cerebral palsy. GMFM-88 is four-point ordinal scale (0-3) with 88 items categorized in to 5 dimensions such as: lying and rolling (17 items), sitting (20 items), crawling and kneeling (14 items), standing (13 items), and walking, running and jumping (24 items). the average score ranges from 0-100. Higher scores indicate better capacity. The GMFM-88 reliability values range from 0.87 to 0.99
Trunk Control Motor Scale (TCMS) | Baseline
  Trunk control motor scale consist of 15 items which are used to assess the sitting balance of trunk control during functional activities such as: (a) while static condition (b) while dynamic condition. TCMS is two, three and four-point ordinal scale with the total score ranges from 0 to 58
Trunk Control Motor Scale (TCMS) | 4th week
  Trunk control motor scale consist of 15 items which are used to assess the sitting balance of trunk control during functional activities such as: (a) while static condition (b) while dynamic condition. TCMS is two, three and four-point ordinal scale with the total score ranges from 0 to 58
Trunk Control Motor Scale (TCMS) | 8th week
  Trunk control motor scale consist of 15 items which are used to assess the sitting balance of trunk control during functional activities such as: (a) while static condition (b) while dynamic condition. TCMS is two, three and four-point ordinal scale with the total score ranges from 0 to 58
Trunk Control Motor Scale (TCMS) | 12th week
  Trunk control motor scale consist of 15 items which are used to assess the sitting balance of trunk control during functional activities such as: (a) while static condition (b) while dynamic condition. TCMS is two, three and four-point ordinal scale with the total score ranges from 0 to 58

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Al-Umeed Rehabilitation Association, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No